CLINICAL TRIAL: NCT02608034
Title: A Two-part, Phase I, Open-label, Multicenter, Two-period, One-sequence Study to Investigate the Effect of Itraconazole and Rifampin on the PK of Vemurafenib at Steady State
Brief Title: A Study to Investigate the Effect of Itraconazole and Rifampin on Pharmacokinetics (PK) of Vemurafenib at Steady State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO29475
Record Dates: First submitted 2015-11-03; First posted 2015-11-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Melanoma, BRAF V600 Mutation Positive
MeSH Terms: conditions — Melanoma | interventions — Itraconazole; Rifampin; Vemurafenib

ARMS (1):
- Part 1: Vemurafenib+Itraconazole (Experimental): Part 1: Participants will receive vemurafenib orally BID up to Day 20 (Period A) followed by vemurafenib orally BID along with itraconazole orally once in the morning from Days 21 to 40 (Period B).\nPart 2: Participants will receive vemurafenib orally BID up to Day 20 (Period A) followed by vemurafenib orally BID along with rifampin orally once in the morning from Days 21 to 40 (Period B).
  Interventions: Drug: Itraconazole; Drug: Rifampin; Drug: Vemurafenib

INTERVENTIONS:
Drug: Itraconazole — Itraconazole will be administered as a 200 mg oral solution QD during Part 1 only for 20 consecutive days.
Drug: Rifampin — Rifampin will be administered as a 600 mg oral solution QD during Part 2 only for 20 consecutive days.
Drug: Vemurafenib — Vemurafenib will be administered in both Part 1 and Part 2 at a dose of 960 mg BID for at least 40 conseutive days.

SUMMARY:
This is a two-part, Phase 1, open-label, multicenter, two-period, one-sequence study to investigate the effect of itraconazole and rifampin on the PK of vemurafenib following multiple 960 milligrams (mg) twice daily (BID) dosing in adult participants with unresectable Stage IIIC or Stage IV metastatic melanoma positive for the BRAF V600 mutation, or other malignant tumor types that harbor a V600-activating mutation of BRAF where the participant has no acceptable standard treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age greater than or equal to (>=) 18 years with either unresectable Stage IIIC or Stage IV metastatic melanoma positive for the BRAF V600 mutation, or other malignant tumor types that harbor a V600-activating mutation of BRAF
* Eastern Cooperative Oncology Group Performance Status 0 to 2
* Life expectancy >=12 weeks
* Adequate hematologic and end organ function obtained within 2 weeks prior to first dose of study drug
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to always use two effective methods of contraception including at least one method with a failure rate of <1% per year during the course of the study and for at least 6 months after completion of study treatment
* Negative serum pregnancy test within 7 days prior to commencement of dosing in women of childbearing potential
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of Study Day 1 of Period A
* Allergy or hypersensitivity to components of the vemurafenib formulation
* Experimental therapy within 4 weeks prior to first dose of study drug treatment on Study Day 1 of Period A
* Major surgical procedure or significant traumatic injury within 14 days prior to first dose of study drug treatment on Study Day 1 of Period A, or anticipation of the need for major surgery during study treatment
* Prior anti-cancer therapy (e.g., biologic or other targeted therapy, chemotherapy) within 28 days (6 weeks for nitrosoureas or mitomycin C, and 14 days for hormonal therapy or kinase inhibitors) before the first dose of study treatment on Study Day 1 of Period A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-05-26 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve From Time 0 to 12 Hours Postdose (AUC0-12) | Period A and B: Pre-morning dose on Day 18, 19, and 20 and 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose on Day 20
Maximum observed concentration (Cmax) | Period A and B: Pre-morning dose on Day 18, 19, and 20 and 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose on Day 20
Time to maximum concentration (Tmax) | Period A and B: Pre-morning dose on Day 18, 19, and 20 and 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose on Day 20

SECONDARY OUTCOMES:
Incidence of adverse events | 28 days after last dose of study treatment (last dose = Day 40)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Mary Crowley Medical Research Center, Dallas, Texas, United States
- Israel (3):
  - Rambam Health Care Campus; Oncology, Haifa
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Tel Aviv Sourasky Medical Center; Pharmacy, Tel Aviv
- Russia (3):
  - Republican Clinical Oncologic Dispensary of Republic Of Tatarstan, Kazan'
  - FSBSI "N. N. Blokhin Russian Cancer Research Center", Moscow
  - St. Petersburg Oncology Hospital, Saint Petersburg
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center; Gastroenterology, Seoul
  - Asan Medical Center; Division of Oncology, Seoul
  - Severance Hospital - Yonsei Uni ; Obstetrics & Gynaecology Dept., Seoul